CLINICAL TRIAL: NCT06669013
Title: A Randomized, Multicenter, Open-label Phase III Study of Dinutuximab Beta With Investigator's Choice of Chemotherapy in Patients Under 18 Years of Age With Bone and Soft Tissue Sarcomas With High Levels of GD2 Expression and Disease Progression During 1st Line Chemotherapy
Brief Title: Chemo-immunotherapy in Patients Under 18 Years of Age With Bone and Soft Tissue Sarcomas
Acronym: FollowTheDIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 821052021
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Bone Sarcoma; Embryonal Rhabdomyosarcoma; Alveolar Rhabdomyosarcoma
MeSH Terms: conditions — Bone Neoplasms; Rhabdomyosarcoma, Embryonal; Rhabdomyosarcoma, Alveolar | interventions — dinutuximab

STUDY DESIGN:
Intervention Model Description: patients with advanced/metastatic GD2-positive rhabdomyosarcoma after progression on 1st line of chemotherapy, advanced/metastatic GD2-positive Ewing sarcoma after progression on 1st line of chemotherapy and advanced/metastatic GD2-positive osteosarcoma after progression on 1st line of chemotherapy.
Who Masked: Participant
Masking Description: Participant Group/Arm
  1. Generalized / metastatic GD2-positive rhabdomyosarcoma after progression on 1st line of chemotherapy.
  2. Generalized / metastatic GD2-positive Ewing sarcoma after progression on 1st line of chemotherapy.
  3. Generalized / metastatic GD2-positive osteosarcoma after progression on 1st line of chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Generalized / metastatic GD2-positive rhabdomyosarcoma (Experimental): Generalized / metastatic GD2-positive rhabdomyosarcoma after progression on 1st line of chemotherapy.
  Chemotherapy options:
  • CARBO(CARBOPLATIN) + ETO(ETOPOSIDE), IFO(IFOSFAMIDE) + ETO(ETOPOSIDE), CARBO(CARBOPLATIN) + IFO(IFOSFAMIDE) (rhabdomyosarcoma)
  + 6 consecutive cycles of dinutuximab beta immunotherapy
  Interventions: Drug: dinutuximab beta
- Generalized / metastatic GD2-positive Ewing sarcoma (Experimental): Generalized / metastatic GD2-positive Ewing sarcoma after progression on 1st line of chemotherapy.
  • ICE (IFOSFAMIDE+CARBOPLATIN+ETOPOSIDE), TEM(TEMOZOLOMIDE+IRINOTECAN), VCT(VINCRISTINE+CYCLOPHOSPHAN+TOPOTECAN), TC(CYCLOPHOSPHAN+TOPOTECAN), TT(TEMOZOLOMIDE+TOPOTECAN), GEM/TAX(GEMCITABINE+DOCETAXEL) (Ewing's sarcoma)
  + 6 consecutive cycles of dinutuximab beta immunotherapy
  Interventions: Drug: dinutuximab beta
- Generalized / metastatic GD2-positive osteosarcoma (Experimental): Generalized / metastatic GD2-positive osteosarcoma after progression on 1st line of chemotherapy.
  • ICE(IFOSFAMIDE+CARBOPLATIN+ETOPOSIDE), IE (IFOSFAMIDE+ETOPOSIDE), CARBOPLATIN+ ETOPOSIDE, Аi(DOXORUBICIN+IFOSFAMIDE), IFO(IFOSFAMIDE), GEM/TAX(GEMCITABINE+DOCETAXEL) (osteosarcoma)
  + 6 consecutive cycles of dinutuximab beta immunotherapy
  Interventions: Drug: dinutuximab beta

INTERVENTIONS:
Drug: dinutuximab beta — Chemotherapy + Immunotherapy (dinutuximab beta)

SUMMARY:
Data from 40 patients are planned to be included in the study to randomize approximately 10 patients.

This study involves patients with advanced/metastatic GD2-positive rhabdomyosarcoma after progression on 1st line of chemotherapy, advanced/metastatic GD2-positive Ewing sarcoma after progression on 1st line of chemotherapy and advanced/metastatic GD2-positive osteosarcoma after progression on 1st line of chemotherapy.

All patients will receive therapy until disease progression (a total of 6 courses of immunotherapy).

The primary objective of the study is to determine the efficacy and safety of dinutuximab beta with investigator's choice of chemotherapy.

DETAILED DESCRIPTION:
Data from 40 patients are planned to be included in the study to randomize approximately 10 patients.

This study involves patients with advanced/metastatic GD2-positive rhabdomyosarcoma after progression on 1st line of chemotherapy, advanced/metastatic GD2-positive Ewing sarcoma after progression on 1st line of chemotherapy and advanced/metastatic GD2-positive osteosarcoma after progression on 1st line of chemotherapy.

6 cycles of treatment with dinutuximab beta are provided in combination with 6-8 cycles of chemotherapy during the induction therapy phase. Switching from one chemotherapy regimen to another is not allowed. Dinutuximab beta should be administered as a slow intravenous infusion through a separate catheter using an infusion pump.

All patients will receive therapy until disease progression (a total of 6 courses of immunotherapy).

Treatment response will be assessed by the investigator after 2, 4 cycles of treatment and at the end of the reinduction therapy period (i.e., after 6 cycles of dinutuximab beta treatment and 6 - 8 cycles of polychemotherapy). Treatment response will be assessed by tumor response according to the criteria for response assessment in the treatment of solid tumors (RECIST 1.1).

After discontinuation of therapy, all patients will be followed up for 6 months. All patients should be followed up to assess survival unless consent is withdrawn. Long-term follow-up/survival assessment visits will be performed monthly until death, withdrawal of consent, or study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form;
2. Age under 18 years of age;
3. Histologically confirmed GD2-positive osteogenic sarcoma, Ewing's sarcoma, soft tissue and undifferentiated sarcomas;
4. Prior to study enrollment, patients must have been treated with one or more lines of adequate chemotherapy and must have relapsed on this therapy or have refractoriness to it;
5. General satisfactory condition of the patient (Lansky scale activity 80-100% (children under 16 years of age), Karnofsky scale 80-100% (children over 16 years of age); ECOG - 0-1);
6. Sufficient cardiopulmonary reserves of the patient's organism (ECG (ELECTROCARDIOGRAPHY) data within normal limits, ventricular ejection fraction > 75% of the upper limit of normal;
7. Adequate liver function (ALT (ALANINE AMINOTRANSFERASE) ≤ 2.5 * VGN, AST (ASPARTATE AMINOTRANSFERASE) ≤ 2.5 * VGN), kidney (creatinine <1.5 * VGN), red bone marrow (granulocytes> 2.0 * 109/L, platelets> 150 * 109/L).

   Six months later, two additional criteria were formulated:
8. Life expectancy at the time of initiation of therapy within the framework of the study is not less than 12 months
9. Oligometastasis disease (presence of 1 to 5 distant metastatic foci) at restaging at the time of the decision to include the patient in the study;

Exclusion Criteria:

1. Withdrawal of consent by the patient or his/her parent/guardian.
2. Exclusion of the patient by the investigator for safety or ethical reasons.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  PFS will be assessed from the date of the first induction dose of dinutuximab beta to the date of first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS will be assessed from the date of administration of the first induction dose of dinutuximab beta to the date of death.
Overall response rate (ORR) | 6 months
  ORR will be assessed by tumor response CR or PR.
Tumor control rate (TCR) | 6 months
  TCR will be assessed by tumor response according CR + PR + stabilization.
Duration of response (DR) | 6 months
  DR will be assessed from initial response to disease progression.
Immune-associated adverse events (IAAE) | 6 months
  IAAE will be assessed from the date of administration of the first induction dose of dinutuximab beta to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Kulyova, MD, Phd, Principal Investigator — Head of Children's Oncology Department
Locations (1):
- Kulyova Svetlana, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No